CLINICAL TRIAL: NCT00438412
Title: Vasoactive Hormones and Oxygen Saturation During Apneic Events in Patients With Obstructive Sleep Apnea
Status: Suspended | Type: Observational
Why Stopped: It was not possible to recruit enough patients with obstructive sleep apnea.
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Pia Holland Gjørup, Department of Medical Research
Other Study IDs: MED.RES.HOS.2006.01.PHH
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Noradrenalin; Endothelin-1; Angiotensin II; Arginine vasopressin; Aldosterone; Renin; Atrial natriuretic peptide; Brain natriuretic peptide; Blood pressure; Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Insipidus; Apnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The mechanisms involved in development and maintenance of hypertension in obstructive sleep apnea are not clarified.

We hypothesize that patients with obstructive sleep apnea have an abnormal level of some vasoactive hormones during apneic events during sleep.

ELIGIBILITY:
Patients with Obstructive sleep apnea

Inclusion Criteria:

* Severe obstructive sleep apnea (apnea-hypopnea index > 30)

Exclusion Criteria:

* Drug or alcohol abuse
* Pregnancy
* History or clinical signs of disease in the heart, lungs, brain, liver, kidneys or endocrine organs
* Diabetes

Healthy Controls

Inclusion Criteria:

* Apnea-hypopnea index < 10

Exclusion criteria:

* Drug or alcohol abuse
* Pregnancy
* History or clinical signs of disease in the heart, lungs, brain, liver, kidneys or endocrine organs
* Diabetes

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults, males and females,age 30 -65
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Regional Hospital Holstebro
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Denmark